CLINICAL TRIAL: NCT06513533
Title: Effect of Dimethyl Fumarate Administered to Patients With Adrenomyeloneuropathy: a Multicenter, Placebo Controlled, Phase IIb/III Trial
Brief Title: Dimethyl Fumarate in Adrenomyeloneuropathy
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Pujol, Aurora, M.D. (Individual)
Collaborators: Instituto de Salud Carlos III (Other Government); Spanish Clinical Research Network - SCReN (Network); Institut d'Investigació Biomèdica de Bellvitge (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: XAMNDMFAP2022; 2021-003826-65 (EudraCT Number)
Record Dates: First submitted 2024-07-17; First posted 2024-07-22 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Adrenomyeloneuropathy Without Cerebral Involvement
MeSH Terms: interventions — Dimethyl Fumarate

STUDY DESIGN:
Intervention Model Description: Double-arm, randomized, placebo-controlled, multicentric trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: Group 1: oral administration of dimethyl fumarate for 36 months Group 2: oral administration of placebo for 24 months, followed by oral dimethyl fumarate for 12 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DMF arm (Experimental): Oral administration of dimethyl fumarate, 480 mg/day, for 36 months
  Interventions: Drug: Dimethyl fumarate
- Placebo arm (Placebo Comparator): Oral administration of placebo for 24 months, followed by oral dimethyl fumarate, 480 mg/day for 12 months
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Placebo — 1 tablet twice daily (one in the morning and one in the evening) for the first 7 days as a starter dose followed by 2 tablets (240 mg) twice daily
  Arms: Placebo arm
Drug: Dimethyl fumarate — 1 tablet twice daily (one in the morning and one in the evening) for the first 7 days as a starter dose followed by 2 tablets (240 mg) twice daily
  Other Names: Skilarence; Tecfidera
  Arms: DMF arm

SUMMARY:
The goal of this clinical trial is to determine if dimethyl fumarate is effective in treating motor problems in adults with Adrenomyeloneuropathy. The trial will also assess the safety of dimethyl fumarate and explore the molecular mechanisms underlying the disease. The primary questions it aims to answer are:

* Does dimethyl fumarate improve motor problems in participants?
* What medical issues do participants experience while taking dimethyl fumarate? Researchers will compare the effects of dimethyl fumarate to a placebo (a substance that looks like the drug but contains no active ingredients) to evaluate its effectiveness in treating Adrenomyeloneuropathy.

Participants will:

* Take either dimethyl fumarate or a placebo daily for 36 months.
* Visit the clinic at the start of the trial, then at 3 months, 6 months, and every 6 months thereafter for checkups and tests.

DETAILED DESCRIPTION:
Adrenoleukodystrophy (X-ALD) is the most prevalent rare genetic disorder affecting the brain's white matter. It is caused by mutations in the ABCD1 gene, which encodes a transporter involved in the degradation of very long-chain fatty acids (VLCFA). As a result, VLCFA accumulate in tissues and plasma, serving as a pathognomonic biomarker for diagnosis. The disease manifests in two main forms: i) adrenomyeloneuropathy (AMN), characterized by chronic progressive spastic paraplegia due to distal axonopathy, and ii) cerebral ALD (cALD), a rapidly progressing and fatal demyelinating leukodystrophy. Current therapeutic options are inadequate, limited to bone marrow transplants and gene therapy for patients with cerebral inflammation. No treatment is available for AMN, which affects 60% of patients.

We have discovered that excess VLCFA leads to mitochondrial reactive oxygen species (ROS) production and oxidative damage, a major factor driving pathogenesis. More recently, we found that the main endogenous response to oxidative damage (the NRF-2 pathway) is impaired in X-ALD. Preclinical tests with an NRF2 activator, specifically the current treatment for multiple sclerosis, dimethyl fumarate (DMF/Tecfidera), showed promising results. All major molecular and cellular pathogenic mechanisms were restored, including: i) mitochondrial function and biogenesis, ii) redox homeostasis, iii) bioenergetic failure, iv) neuroinflammation, along with axonal damage and clinical signs of the disease such as locomotor disability. Consequently, we obtained an international patent for repurposing DMF for X-ALD (US15/957,601) and Orphan Drug Designation by the EMA in 2020 (EMA/OD/0000010028).

Now we are translating this knowledge into a randomized phase IIb/III double-blind placebo-controlled study over 36 months for 40 AMN patients, to determine if DMF is effective in these patients. For the first 24 months, patients will be divided into two groups (placebo and active treatment) in a ratio of 1:2. A 12-month extension phase will follow, during which all patients will receive treatment. Furthermore, we aim to elucidate the molecular mechanisms driving the disease and dissect the redox-inflammatory effects of DMF using an integrative multi-omics approach, which will involve single-cell RNA sequencing in PBMC, and lipidomics in plasma. The clinical and molecular data from historical national and international AMN and cALD cohorts will be pooled to identify markers of severity and progression. Our goal is to address unmet needs in AMN while generating novel fundamental knowledge that will be useful for this and other common axonopathies.

ELIGIBILITY:
Inclusion Criteria:

* Men and women of 18 to 65 years old at the time of the inclusion, suffering from AMN with:

  * elevated plasma VLCFA
  * ABCD1 gene mutation identified
* Clinical signs of AMN with at least pyramidal signs in the lower limbs and difficulties to walk (EDSS score ≥ 2.0 and ≤ 6.5). EDSS score will also be re-evaluated at M12, M24 and M36.
* Normal brain MRI or brain MRI showing:

  * abnormalities that can be observed in AMN patients without cerebral demyelination with a maximum Loes score of 4
  * and/or stable (≥ 6 months) cerebral demyelination without gadolinium enhancement with a Loes score ≤ 12
* Appropriate steroid replacement if adrenal insufficiency is present
* Potential childbearing women should use an adequate method of contraception to avoid pregnancy throughout the study to minimize the risk of pregnancy. If oral contraceptives are used, the use of an alternative barrier method is recommended.
* Likely to be able to participate in all scheduled evaluations and complete all required study procedures
* Signed and dated written informed consent to participate in the study in accordance with local regulations

Exclusion Criteria:

* Any progressive neurological disease other than AMN
* Leukopenia below 3.0x109/L, lymphopenia below 0.5x109/L or other pathological results in the complete blood count
* Suspected or confirmed progressive multifocal leukoencephalopathy (PML)
* Severe gastrointestinal disease
* Uncontrolled hepatic, renal or cardiovascular disease, or any evolutive malignancy
* Pregnancy and breast-feeding in woman and potential childbearing woman unable or unwilling to use an acceptable contraceptive method during the study
* Any new medication for AMN initiated less than three months prior to inclusion
* Contra-indications for MRI procedure such as subjects with paramagnetic materials in the body as aneurysm clips, pacemakers, intraocular metal or cochlear implants
* Inclusion in another therapeutic clinical trial for ALD
* Not easily contactable by the investigator in case of emergency or not able to call the investigator

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-04-23 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Postural sway test | Interim analysis 1 (at 12 months of treatment)
  Balance is assessed with static posturography by measuring the extent of postural sway in four conditions, each for two 20-second trials: (1) eyes open feet shoulder width apart (EOFA), (2) eyes closed feet shoulder width apart (ECFA), (3) eyes open feet together (EOFT), and (4) eyes closed feet together (ECFT)
Postural sway test | Final analysis 1 (at 24 months of treatment)
  Balance is assessed with static posturography by measuring the extent of postural sway in four conditions, each for two 20-second trials: (1) eyes open feet shoulder width apart (EOFA), (2) eyes closed feet shoulder width apart (ECFA), (3) eyes open feet together (EOFT), and (4) eyes closed feet together (ECFT)
Postural sway test | Final analysis 2 (at 36 months of treatment)
  Balance is assessed with static posturography by measuring the extent of postural sway in four conditions, each for two 20-second trials: (1) eyes open feet shoulder width apart (EOFA), (2) eyes closed feet shoulder width apart (ECFA), (3) eyes open feet together (EOFT), and (4) eyes closed feet together (ECFT)

SECONDARY OUTCOMES:
2 Minute Walk Test (2MWT) | Interim analysis 1 (at 6 months of treatment)
  It measures the distance an individual is able to walk over a total of two minutes on a hard, flat surface.
2 Minute Walk Test (2MWT) | Interim analysis 2 (at 12 months of treatment)
  It measures the distance an individual is able to walk over a total of two minutes on a hard, flat surface.
2 Minute Walk Test (2MWT) | Final analysis 1 (at 24 months of treatment)
  It measures the distance an individual is able to walk over a total of two minutes on a hard, flat surface.
2 Minute Walk Test (2MWT) | Final analysis 2 (at 36 months of treatment)
  It measures the distance an individual is able to walk over a total of two minutes on a hard, flat surface.
6 Minute Walk Test (6MWT) | Interim analysis 1 (at 6 months of treatment)
  It measures the distance an individual is able to walk over a total of six minutes on a hard, flat surface
6 Minute Walk Test (6MWT) | Interim analysis 2 (at 12 months of treatment)
  It measures the distance an individual is able to walk over a total of six minutes on a hard, flat surface
6 Minute Walk Test (6MWT) | Final analysis 1 (at 24 months of treatment)
  It measures the distance an individual is able to walk over a total of six minutes on a hard, flat surface
6 Minute Walk Test (6MWT) | Final analysis 2 (at 36 months of treatment)
  It measures the distance an individual is able to walk over a total of six minutes on a hard, flat surface
Time to walk 25 Feet (TW25) | Interim analysis 1 (at 6 months of treatment)
  The TW25 (time to walk 25 feet) is a widely used outcome measure of Leg function/ambulation
Time to walk 25 Feet (TW25) | Interim analysis 2 (at 12 months of treatment)
  The TW25 (time to walk 25 feet) is a widely used outcome measure of Leg function/ambulation
Time to walk 25 Feet (TW25) | Final analysis 1 (at 24 months of treatment)
  The TW25 (time to walk 25 feet) is a widely used outcome measure of Leg function/ambulation
Time to walk 25 Feet (TW25) | Final analysis 2 (at 36 months of treatment)
  The TW25 (time to walk 25 feet) is a widely used outcome measure of Leg function/ambulation
Stair-climbing | Interim analysis 1 (at 12 months of treatment)
  Participants are timed using a hand-held stopwatch as they ascended one flight of 4 steps as quickly and safely as possible with handrail use allowed as needed
Stair-climbing | Final analysis 1 (at 24 months of treatment)
  Participants are timed using a hand-held stopwatch as they ascended one flight of 4 steps as quickly and safely as possible with handrail use allowed as needed
Stair-climbing | Final analysis 2 (at 36 months of treatment)
  Participants are timed using a hand-held stopwatch as they ascended one flight of 4 steps as quickly and safely as possible with handrail use allowed as needed
Strength | Interim analysis 1 (at 12 months of treatment)
  The average of two maximal effort break test trials for each side and muscle group is measured using a dynamometer and documented in Kg
Strength | Final analysis 1 (at 24 months of treatment)
  The average of two maximal effort break test trials for each side and muscle group is measured using a dynamometer and documented in Kg
Strength | Final analysis 2 (at 36 months of treatment)
  The average of two maximal effort break test trials for each side and muscle group is measured using a dynamometer and documented in Kg
SF-Qualiveen (Short-Form Qualiveen) | Interim analysis 1 (at 12 months of treatment)
  The Qualiveen is a specific patients' health-related quality of life developed to assess the impact of urinary disorders in patients with neurological conditions.
SF-Qualiveen (Short-Form Qualiveen) | Final analysis 1 (at 24 months of treatment)
  The Qualiveen is a specific patients' health-related quality of life developed to assess the impact of urinary disorders in patients with neurological conditions.
SF-Qualiveen (Short-Form Qualiveen) | Final analysis 2 (at 36 months of treatment)
  The Qualiveen is a specific patients' health-related quality of life developed to assess the impact of urinary disorders in patients with neurological conditions.
Revised Fecal Incontinence Scale (RFIS) | Interim analysis 1 (at 12 months of treatment)
  The RFIS is a short, reliable, and valid five item scale that can be used to assess fecal incontinence and to monitor patient outcomes following treatment.
Revised Fecal Incontinence Scale (RFIS) | Final analysis 1 (at 24 months of treatment)
  The RFIS is a short, reliable, and valid five item scale that can be used to assess fecal incontinence and to monitor patient outcomes following treatment.
Revised Fecal Incontinence Scale (RFIS) | Final analysis 2 (at 36 months of treatment)
  The RFIS is a short, reliable, and valid five item scale that can be used to assess fecal incontinence and to monitor patient outcomes following treatment.
Brain neuroimaging: Loes | Interim analysis 1 (at 12 months of treatment)
  The Loes score is a 34-point imaging-based severity scale-based scoring system for patients with X-ALD based on the neuroanatomical involvement and the presence or absence of total and/or global atrophy. This 34-point imaging-based severity scale was based on the location and extent of central nervous system involvement and presence of either focal or global atrophy.
Brain neuroimaging: Loes | Final analysis 1 (at 24 months of treatment)
  The Loes score is a 34-point imaging-based severity scale-based scoring system for patients with X-ALD based on the neuroanatomical involvement and the presence or absence of total and/or global atrophy. This 34-point imaging-based severity scale was based on the location and extent of central nervous system involvement and presence of either focal or global atrophy.
Brain neuroimaging: Loes | Final analysis 2 (at 36 months of treatment)
  The Loes score is a 34-point imaging-based severity scale-based scoring system for patients with X-ALD based on the neuroanatomical involvement and the presence or absence of total and/or global atrophy. This 34-point imaging-based severity scale was based on the location and extent of central nervous system involvement and presence of either focal or global atrophy.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Casasnovas, MD, PhD, Principal Investigator — Bellvitge University Hospital
Locations (3):
- Spain (3):
  - Bellvitge University Hospital, L'Hospitalet de Llobregat, Barcelona
  - Donostia University Hospital, Donostia / San Sebastian
  - University Hospital 12 de Octubre, Madrid

IPD SHARING:
Plan to Share IPD: No